CLINICAL TRIAL: NCT01436214
Title: Phase 1/2a, Open-Label, Dose-Escalation and Safety Study of APC-100 [Pentamethylchromanol, 2,2,5,7,8-Pentamethyl-6] in Men With Advanced Prostate Cancer
Brief Title: Dose-Escalation and Safety Study of APC-100 for the Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adamis Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APC-100-01
Record Dates: First submitted 2011-08-31; First posted 2011-09-19 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APC-100 (Experimental)
  Interventions: Drug: APC-100

INTERVENTIONS:
Drug: APC-100 — Daily oral, dose escalation, 28-day cycle(s)

SUMMARY:
This study is a phase 1/2a, open label, dose escalation and safety study of APC-100 (2,2,5,7,8-Pentamethyl-6-chromanol) in men with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically proven adenocarcinoma of the prostate
* Patients must have progressive disease
* Patients must have had prior treatment with bilateral orchiectomy or androgen deprivation therapy with an LHRH-blocker with evidence of treatment failure

Exclusion Criteria:

* Patients treated with other secondary hormonal therapies
* Patients with prior chemotherapy given for castrate-resistant prostate cancer
* Patients with prior radiation therapy completed less than 4 weeks prior enrollment
* Patients with prior investigational therapies within 4 weeks before treatment with APC-100
* Evidence of active second malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and recommended Phase 2a Dose | Within 12 weeks following treatment
  Determination of the MTD based on documentation of dose-limiting toxicities (DLTs) and adverse events. Eighteen patients will be accrued for this part of the study. The MTD will be determined based on both the acute DLTs (within the first cycle of treatment) and late (within cycles 2 through 3) DLTs of APC-100. The establishment of a recommended phase 2a dose will be based on toxicity (DLTs within the first 28 days) and tolerability (DLTs within the first 12 weeks) of APC-100.

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) profile of APC-100 | Pre-Dose, Cycle 1:Day 1, Cycle 2:Day 2,Pre-Dose on Day 1 of each additional cycle
  Single dose and steady state pharmacokinetics of APC-100 by oral administration daily for 28 consecutive days on a 28-day cycle will be determined. The following PK parameters (half-life, Cmax, Tmax, AUC, CI, CIr and V) will be determined.
Assess number, types, and severity of toxicity and adverse events | 12 weeks
  Assessment of incidence, severity, duration, causality and types of toxicity and adverse event severities assessed by NCI Common Toxicity Criteria (NCI CTC), version 4.0)
Assess preliminary evidence of anti-tumor activity through PSA response | pre-study, Cycle 1: Day 1 (unless prestudy was performed within 7 days of study entry), Cycle 2: Day 1, End of Treatment
  Assessment of preliminary anti-tumor activity will be based on PSA response (absolute and percentage change compared to prestudy (baseline) and RECIST criteria, if the patient has measurable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I Heath, MD, Principal Investigator — Wayne State University; Jeremy Cetnar, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin